CLINICAL TRIAL: NCT01307917
Title: Endothelial Dysfunction and the Role of Flavonoids in the Prevention of Nephropathy Among Pediatric Patients With Diabetes
Brief Title: Flavonoids in the Treatment of Endothelial Dysfunction in Children With Diabetes
Acronym: flavonoid
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding ever received
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A09-3502
Record Dates: First submitted 2010-11-15; First posted 2011-03-03 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Diabetic Nephropathy; Endothelial Dysfunction
Keywords: diabetes mellitus; diabetic nephropathy; vascular endothelial dysfunction; flavonoids; flow-mediated dilation
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus | interventions — Flavonoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- healthy controls high flavonoid (Experimental): 20 healthy adolescents (12-21 years old) receiving the flavonoid-rich capsule/supplement
  Interventions: Dietary Supplement: flavonoids
- healthy controls low flavonoid (Active Comparator): 20 healthy adolescents (12-21 years old) receiving the placebo
  Interventions: Dietary Supplement: flavonoids
- T1DM or T2DM high flavonoid (Experimental): 20 adolescents (12-21 years old) with Type 1 diabetes mellitus or Type 2 diabetes mellitus receiving the capsule/supplement
  Interventions: Dietary Supplement: flavonoids
- T1DM or T2DM low flavonoid (Active Comparator): 20 adolescents (12-21 years old) with Type 1 diabetes mellitus or Type 2 diabetes mellitus receiving the placebo
  Interventions: Dietary Supplement: flavonoids

INTERVENTIONS:
Dietary Supplement: flavonoids — for 14 days, one dose two times per day, subjects will ingest a flavonoid-rich capsule containing 500 mg flavonoids or a placebo capsule made, stored, and dispensed by TTUHSC Pharmacy, with a similar look and taste.

SUMMARY:
Diabetes is the most common metabolic disease of childhood. Vascular disease is a leading complication of diabetes, and attempts to maintain close glycemic control do not prevent the sequelae that claim the lives and quality of life of millions of diabetics each year. Up to forty percent of patients with diabetes mellitus ultimately develop diabetic nephropathy, the most common cause of end-stage renal disease requiring dialysis in the US. Flavonoid-rich diets are a promising intervention to prevent the endothelial dysfunction that apparently leads to this deadly complication. The mechanisms are still unclear but probably involve nitric oxide synthesis. The investigators hypothesize that early maintenance of the integrity of renal vasculature will significantly improve the lifelong prognosis for patients with diabetes. Flavonoids with anti-inflammatory and antioxidant activities could be used to protect endothelial function, and together with good glycemic control, prevent the development and progression of nephropathy. The investigators aims are to:

1. compare endothelial function by studying reactive hyperemia, nitric oxide, and proinflammatory factors in adolescents (12-21 years old) with diabetes versus healthy sex- and age-matched control subjects.
2. identify early markers in urine for vascular endothelial injury.
3. examine the effects of flavonoids on vascular function, urine nitric oxide, and proinflammatory factors in patients with diabetes mellitus.

DETAILED DESCRIPTION:
Our proposal is the first attempt to use flavonoids to treat endothelial dysfunction as a causative factor of nephropathy in a pediatric population with diabetes. The investigators plan to recruit 40 adolescents with type 1 or 2 diabetes mellitus and 40 healthy peers into a double-blind, randomized, controlled study. Peripheral arterial tonometry, a noninvasive method to assess vascular status, will be employed to study endothelial function in both groups. Measurements of renal nitric oxide synthesis will be assayed using a nitric oxide chemiluminescence analyzer. Urinary protein microarray analyses will be conducted to assess early markers of kidney inflammation. The array is a multiplex sandwich fluorescent immunoassay for the simultaneous quantification of interleukin-1b (IL-1b), IL-2, IL-4, IL-6, IL-8, IL-10, IL-12, interferon gamma, tumor necrosis factor-alpha, macrophage inflammatory protein-1-alpha and beta, and RANTES. The initial acute response and effect of 14 days of treatment with a flavonoid-rich capsulated supplement will be compared to a placebo. Study subjects will return for baseline assessments a week after the final flavonoid supplement to evaluate the sustainability of the response. Differences between group means for the measured variables before, during, and after the interventions will be tested for statistical significance using paired t-tests and nonparametric statistics. Univariate correlations will be calculated using Pearson's r.

ELIGIBILITY:
Inclusion Criteria:

* adolescents 12 - 21 years old
* with T1DM or T2DM and their healthy age- and sex-matched peers
* DM subjects must maintain good glycemic control with HbA1C < 11

Exclusion Criteria:

* no co-morbidities that could lead to inflammation or decline in renal function will be allowed
* no non-steroidal anti-inflammatory drugs should be taken, for any reason, within 48 hours prior to the study days
* no smoking will be permitted on the day of Pre-Study Evaluation or Study Days 0, 14, or 21
* controls should not be taking any medications

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
compare endothelial function by studying reactive hyperemia, nitric oxide, and proinflammatory factors in adolescents (12-21 years old) with diabetes vs. healthy sex- and age-matched control subjects. | day 0; day 14; day 21

SECONDARY OUTCOMES:
identify early markers in urine for vascular endothelial injury | screening, day 0, day 14, day 21
examine the effects of flavonoids on vascular function, urine nitric oxide, and proinflammatory factors in patients with diabetes mellitus | day 0, day 14, day 21

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Vasylyeva, MD, PhD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas, United States